CLINICAL TRIAL: NCT06784687
Title: Evaluation of the Prevalence and Clinical Manifestation of SARS-CoV-2 Infection in a Population of Adult and Pediatric Patients With Congenital Heart Disease Not Treated Surgically, and in a Population of Pediatric Patients With Cardiomyopathy, Arrhythmic Pathology, or Pulmonary Hypertension
Brief Title: Evaluation of the Prevalence and Clinical Manifestation of SARS-CoV-2 Infection in a Population of Adult and Pediatric Patients With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIOPEDCOVID
Record Dates: First submitted 2024-12-30; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-11

CONDITIONS: Congenital Heart Disease; Cardiomyopathy; Pulmonary Arterial Hypertension; SARS CoV-2 Infection
MeSH Terms: conditions — Heart Defects, Congenital; Cardiomyopathies; Pulmonary Arterial Hypertension; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study, drug-free, cross-sectional, single-center is to describe the incidence and characteristics of the clinical course and any short- and medium-term complications of patients with congenital heart disease of medical interest, and pediatric patients with cardiomyopathy, arrhythmic pathology or pulmonary arterial hypertension who have been affected by Sars-Cov-2 disease. The secondary objective of the study is to identify risk factors for the development of moderate-severe forms of COVID-19 disease in the study population.

DETAILED DESCRIPTION:
This is an observational, drug-free, cross-sectional, single-centre study. All patients followed at our centre and suffering from congenital heart disease treated with only haemodynamic procedures haemodynamic procedures alone, as well as paediatric patients suffering from cardiomyopathy, pulmonary hypertension or arrhythmic pathology whose follow-up was still in progress at the time of the start of the pandemic (due to death or for reasonsof the patient). The structural collection of data necessary for the evaluation of targets will take place through the creation of a specific electronic archive, in which census of all patients who have undergone follow-up at our centre since 01/01/2005 at the time of study approval and still in follow-up at the time of the start of the pandemic.

Patients of all ages will be enrolled age, both paediatric and adult, followed at our centre. It is estimated to include in the study approximately 5000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages with congenital heart disease undergoing hemodynamic procedures at our center or in natural history
* Pediatric patients with cardiomyopathy, arrhythmic disease, or hypertension pulmonary
* Obtaining informed consent
* Patients who have access to an e-mail address and a computer to complete the questionnaire

Exclusion Criteria:

* Patients with congenital heart disease undergoing corrective or palliative surgical treatment

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients followed at our center and suffering from congenital heart disease treated by hemodynamic procedures alone, as well as pediatric patients with cardiomyopathy, pulmonary hypertension, or arrhythmic disease whose follow-up was still ongoing at the time of the onset of the pandemic
Sampling Method: Non-Probability Sample
Enrollment: 2376 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Severity of SARS-CoV-2 infection evaluation | Upon completion of the questionnaire by patient on day 1
  The presence of ongoing SARS-CoV-2 infection will be defined as detection of viral RNA to a molecular swab or the detection of specific antigen at an antigenic swab, while the presence of previous infection will be defined as the presence of seroconversion for SARS-CoV-2 at a quantitative serological test. Severity of SARS-CoV-2 infection will be defined at different forms:
  * Severe form: Admission to intensive care unit, need for invasive respiratory support, death
  * Moderate form: Need for hospitalization or home oxygen therapy, or Worsening of oxygen dependence in patients on chronic home oxygen therapy.
  * Mild form: Symptomatic patients who do not meet the criteria for moderate or severe disease.
  * Asymptomatic form: Patients with infection positivity who do not have symptoms of disease.
  The patients' medical history and clinical data, as reported in the questionnaire, will be evaluated to look for possible risk factors for the development of severe forms of COVID-19 disease.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Bonetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy